CLINICAL TRIAL: NCT01184430
Title: Monocentric Pilot Study of Effect of Perioperative Hemodynamic Optimization on the Immune Function Parameters of Peripheral Blood Monocytes After Cardiac Surgery
Brief Title: Effect of Perioperative Hemodynamic Optimization on the Immune Function Parameters of Peripheral Blood Monocytes After Cardiac Surgery
Acronym: Algebra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Sander, Vice Chair, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Algebra
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Wound Infection; Postoperative Outcome
Keywords: advanced hemodynamic monitoring; goal-directed therapy; cardiac surgery; hemodynamic monitoring
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- advanced hemodynamic monitoring (Active Comparator): advanced hemodynamic monitoring with pulse contour analysis ( LiDCO rapid) and goal-directed therapy
  Interventions: Device: Pulse contour cardiac output device
- standard monitoring (No Intervention): hemodynamic monitoring based on the standard operating procedures of our clinic

INTERVENTIONS:
Device: Pulse contour cardiac output device — Goal directed volume therapy using stroke volume variation and cardiac output to guide volume therapy and inotropic support.
  Other Names: Non calibrated pulse contour cardiac output monitor
  Arms: advanced hemodynamic monitoring

SUMMARY:
Cardiac surgery patients have a high risk to suffer from postoperative infections. Some studies have shown, that humoral and cellular factors are associated with perioperative immunodysfunction and can increase the risk of postoperative infections. Monocytes in the blood and, especially alveolar macrophages are important for an adequate host defence. In studies the investigators have shown that hemodynamic parameters have a significant influence on the probability to develop postoperative infections. The aim of the study is to investigate, whether cardiac surgery patients have an altered immune function after surgery that is predictive for the latter development of subsequent infections and whether they benefit from a goal-directed volume and hemodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery patient undergoing cardiopulmonary bypass
* signed informed consent

Exclusion Criteria:

* pregnant or breast feeding women
* Age <18 years
* pulmonary disease with an oxygenation index <300mmHg
* liver disease (>Child B)
* HIV-Infection
* Therapy with corticosteroids
* Condition after transplantation
* preexisting infection before operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
HLA-DR Expression on monocytes after surgery | 24 hours

SECONDARY OUTCOMES:
ICU stay | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, MD, Principal Investigator — Dept. of Anesthesiology Charité Universitaetsmedizin Berlin; Claudia Spies, MD, Study Chair — Dept. of Anesthesiology Charité Universitaetsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum, Berlin, Germany